CLINICAL TRIAL: NCT05889182
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate Efficacy and Safety of Upadacitinib in Adult and Adolescent Subjects With Moderate to Severe Hidradenitis Suppurativa Who Have Failed Anti-TNF Therapy
Brief Title: A Study to Assess Change in Disease Activity and Adverse Events of Oral Upadacitinib in Adult and Adolescent Participants With Moderate to Severe Hidradenitis Suppurativa Who Have Failed Anti-TNF Therapy
Acronym: Step-Up HS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-698; 2023-503661-28-00 (Other: EU CT)
Record Dates: First submitted 2023-05-26; First posted 2023-06-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Upadacitinib; ABT-494; Rinvoq; STEP-UP HS
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Period 1: Upadacitinib Dose A (Experimental): Participants will receive Upadicitinib Dose A once daily for 16 weeks.
  Interventions: Drug: Upadacitinib
- Period 1: Placebo (Placebo Comparator): Participants will receive Placebo once daily for 16 weeks.
  Interventions: Drug: Placebo
- Period 2: Group 1 - Upadacitinib Dose A (Experimental): Participants who were randomized to placebo in Period 1 who did not achieve HiSCR 50 (clinical non-responder, CNR) at Week 16 will receive Upadacitinib Dose A once daily for 20 weeks.
  Interventions: Drug: Upadacitinib
- Period 2: Group 2 - Placebo (Placebo Comparator): Participants who were randomized to placebo in Period 1 who achieve HiSCR 50 (clinical responder, CR) at Week 16 will continue to receive placebo once daily for 20 weeks.
  Interventions: Drug: Placebo
- Period 2: Group 3 - Upadacitinib Dose A (Experimental): Participants who were randomized to upadacitinib Dose A in Period 1 who did not achieve HiSCR 50 (CNR) at Week 16 will continue to receive upadacitinib Dose A once daily for 20 weeks.
  Interventions: Drug: Upadacitinib
- Period 2: Group 4 - Upadacitinib Dose A (Experimental): Participants who were randomized to upadacitinib Dose A in Period 1 who achieve HiSCR 50 (CR) at Week 16 will receive upadacitinib Dose A once daily for 20 weeks.
  Interventions: Drug: Upadacitinib
- Period 2: Group 5 - Upadacitinib Dose B (Experimental): Participants who were randomized to upadacitinib Dose A in Period 1 who achieve HiSCR 50 (CR) at Week 16 will receive upadacitinib Dose B once daily for 20 weeks.
  Interventions: Drug: Upadacitinib
- Period 2: Group 6 - Placebo (Experimental): Participants who were randomized to upadacitinib Dose A in Period 1 who achieve HiSCR 50 (CR) at Week 16 will receive placebo once daily for 20 weeks.
  Interventions: Drug: Placebo
- Period 3: Long-Term Extension (Experimental): Eligible participants will continue to receive upadacitinib or placebo for 68 weeks. Participants will be followed-up for approximately 30 days.
  Interventions: Drug: Upadacitinib; Drug: Placebo

INTERVENTIONS:
Drug: Upadacitinib — Oral Tablets
  Other Names: ABT-494; RINVOQ
  Arms: Period 1: Upadacitinib Dose A; Period 2: Group 1 - Upadacitinib Dose A; Period 2: Group 3 - Upadacitinib Dose A; Period 2: Group 4 - Upadacitinib Dose A; Period 2: Group 5 - Upadacitinib Dose B; Period 3: Long-Term Extension
Drug: Placebo — Oral Tablets
  Arms: Period 1: Placebo; Period 2: Group 2 - Placebo; Period 2: Group 6 - Placebo; Period 3: Long-Term Extension

SUMMARY:
Hidradenitis suppurativa (HS) is an inflammatory skin disease that causes painful lesions in the axilla (underarm), inguinal (groin) and anogenital (anal/genital) regions. This study will assess how safe and effective upadacitinib is in treating adult and adolescent participants with moderate to severe HS who have failed to respond to or are intolerant of anti-tumor necrosis factor (TNF) therapy. Adverse events and change in disease activity will be assessed.

Upadacitinib is an approved drug for ulcerative colitis, atopic dermatitis, rheumatoid arthritis, psoriatic arthritis, and axial spondylarthritis and is being developed for the treatment of HS. This study is "double-blinded", meaning that neither the trial participants nor the study doctors will know who will be given upadacitinib and who will be given placebo. This study is comprised of 3 periods. In Period 1, participants are randomized into 2 groups called treatment arms where each group receives a different treatment. There is a 1 in 2 chance that participants will be assigned to placebo. In Period 2, participants are placed into 6 different groups depending on their placement and results in Period 1. Period 3 is the long-term extension period where participants will continue treatment from Period 2. Approximately 1328 adult and adolescent participants diagnosed with HS will be enrolled in approximately 300 sites worldwide.

Participants will receive oral tablets of upadacitinib or placebo once daily for 36 weeks in Period 1 and Period 2. Eligible participants from Period 1 and Period 2 will enter Period 3 and receive oral tablets of upadacitinib or placebo once daily for 68 weeks. Participants will be followed up for approximately 30 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular outpatient visits during the study. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hidradenitis suppurativa (HS) for at least 6 months prior to Baseline, as determined by the investigator (i.e., through medical history and interview of participant).
* Documented history of previous use of >= 1 tumor necrosis factor (TNF) inhibitor for HS for at least 12 weeks and/or 1 approved non-anti-TNF biologic therapy for HS for at least 16 weeks characterized by inadequate response or for any duration characterized by intolerance as determined by the investigator.
* Participant must have a total abscess and inflammatory nodule (AN) count of >= 5 at Baseline.
* HS lesions must be present in at least 2 distinct anatomic areas at Baseline.
* At least 1 anatomic area of HS involvement characterized as Hurley Stage II or higher at Baseline.
* Draining fistula count of <= 20 at Baseline.

Exclusion Criteria:

* History of active skin disease other than HS that could interfere with the assessment of HS, including skin infections (bacterial, fungal, or viral) requiring systemic treatment within 4 weeks of the Baseline visit.
* Treatment with any investigational drug of chemical or biologic nature within a minimum of 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug or be currently enrolled in another interventional clinical study. Investigational drugs are also prohibited during the study.
* Previous treatment with any cell-depleting therapies including but not limited to anti-CD20 (e.g., rituximab) within 12 months prior to Baseline or until B cell count returns to normal level or pre-treatment level.
* Use of prescription topical therapies (including topical antibiotics) that can also be used to treat HS within 14 days prior to the Baseline visit.
* Received any systemic (including oral) antibiotic treatment for HS or any other chronic inflammatory disorder within 14 days prior to the Baseline visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1328 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Hidradenitis Suppurative Clinical Response (HiSCR) 50 | Baseline to Week 16
  HiSCR 50 is defined as at least a 50% reduction in the total abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to Baseline.
Number of Participants with Adverse Events (AEs) | Up to Approximately Week 108
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change from Baseline in Draining Fistula Count | Baseline to Week 16
  Change from baseline in draining fistula count.
Percentage of Participants Achieving Hidradenitis Suppurative Clinical Response (HiSCR) 75 | Baseline to Week 16
  HiSCR 75 is defined as at least a 75% reduction in the total abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to Baseline.
Percentage of Participants Achieving Numeric Rating Scale 30 (NRS30) at Week 4 Among Participants with NRS ≥ 3 at Baseline | Baseline to Week 4
  Achievement will be considered at least a 30% reduction and at least 2 units reduction from Baseline in the Participant's Global Assessment (PGA) of HS-related skin pain NRS based on worst skin pain in a 24-hour recall period (maximal daily pain). The PGA Skin Pain is an 11-point numerical rating scale with ratings for the item ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine).
Change from Baseline in Hidradenitis Suppurativa Symptom Assessment (HSSA) | Baseline to Week 16
  The HSSA (24-hour recall) is a 9-item PRO questionnaire developed to assess the primary symptoms of HS in the 7 consecutive days prior to assessments. Each item of the HSSA is scored on an 11-point (0 to 10) NRS, where 0 represents no symptoms and 10 represents extreme symptom experience.
Change from Baseline in Hidradenitis Suppurativa Impact Assessment (HSIA) | Baseline to Week 16
  The HSIA is an 18-item PRO questionnaire developed to assess the impact of HS on the daily lives of subjects in the 7 days prior to the assessment. Items 1 - 16 of the HSIA are scored on a 0 to 10 NRS, where 0 represents no impact and 10 represents extreme impact.
Change from Baseline in Dermatology Life Quality Index (DLQI) for Adult Participants and Adolescent Participants Age ≥16 Years Old and Older | Baseline to Week 16
  The DLQI and the CDLQI are both 10-item questionnaires used to assess the impact of hidradenitis suppurativa (HS) disease symptoms and treatment on quality of life that consists of 10 questions scored on a 4-point scale where 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much.
Change from Baseline in Hidradenitis Suppurativa (HS)-Related Odor, Based on Hidradenitis Suppurativa Symptom Assessment (HSSA) Question 8 | Baseline to Week 16
  The HSSA (24-hour recall) is a 9-item PRO questionnaire developed to assess the primary symptoms of HS in the 7 consecutive days prior to assessments. Each item of the HSSA is scored on an 11-point (0 to 10) NRS, where 0 represents no symptoms and 10 represents extreme symptom experience.
Change from Baseline in the Patient's Global Assessment of Hidradenitis Suppurativa (HS)-Related Skin Pain NRS | Baseline to Week 8
  The PGA Skin Pain is an 11-point numerical rating scale with ratings for the item ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine) that is used to assess the worst pain due to HS. Patients are asked to respond to the item based on a recall period of "the last 24 hours
Occurrence of Hidradenitis Suppurativa (HS) Flare During Period 1 | Baseline to Week 16
  Defined as at least one occurrence of a ≥ 25% increase in AN count, with a minimum absolute increase of 2 relative to Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (285):
- United States (87):
  - Cahaba Dermatology & Skin Health Center /ID# 254876, Birmingham, Alabama
  - Peak Dermatology Aesthetics and Wellness Fountain Hills /ID# 272564, Fountain Hills, Arizona
  - Medical Dermatology Specialists /ID# 254226, Phoenix, Arizona
  - Mayo Clinic - Scottsdale /ID# 254388, Scottsdale, Arizona
  - Banner University Medicine Dermatology /ID# 255853, Tucson, Arizona
  - Clinical Trials Institute - Northwest Arkansas /ID# 254924, Fayetteville, Arkansas
  - Burke Pharmaceutical Research /ID# 254238, Hot Springs, Arkansas
  - Arkansas Research Trials /ID# 254233, North Little Rock, Arkansas
  - NW Arkansas Clinical Trials Center /ID# 254311, Rogers, Arkansas
  - Private Practice - Dr. Tooraj Raoof /ID# 254374, Encino, California
  - Marvel Clinical Research /ID# 276228, Huntington Beach, California
  - Dermatology Research Associates /ID# 254846, Los Angeles, California
  - NorCal Clinical Research /ID# 274219, Rocklin, California
  - Integrative Skin Science and Research /ID# 254930, Sacramento, California
  - University of California Davis Health /ID# 254229, Sacramento, California
  - Medderm Associates /ID# 253800, San Diego, California
  - Clinical Trials Research Institute /ID# 254466, Thousand Oaks, California
  - UConn Health Main /ID# 254507, Farmington, Connecticut
  - Yale University School of Medicine /ID# 254586, New Haven, Connecticut
  - Skin Care Research Boca Raton /ID# 253814, Boca Raton, Florida
  - Apex Clinical Trials /ID# 255756, Brandon, Florida
  - Florida Academic Dermatology Center /ID# 254011, Coral Gables, Florida
  - Dermatology Associates of the Palm Beaches /ID# 275950, Delray Beach, Florida
  - Skin Care Research - Hollywood /ID# 254508, Hollywood, Florida
  - Life Clinical Trials /ID# 258613, Margate, Florida
  - Skin Care Research - Tampa /ID# 256440, Tampa, Florida
  - Advanced Clinical Research Institute /ID# 253746, Tampa, Florida
  - Avita Clinical Research /ID# 254471, Tampa, Florida
  - Centricity Research /ID# 255470, Columbus, Georgia
  - Treasure Valley Medical Research /ID# 255208, Boise, Idaho
  - DeNova Research /ID# 254372, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine /ID# 254503, Chicago, Illinois
  - NorthShore University HealthSystem - Skokie /ID# 254389, Skokie, Illinois
  - Dawes Fretzin, LLC /ID# 254390, Indianapolis, Indiana
  - Options Research Group /ID# 254537, West Lafayette, Indiana
  - U.S. Dermatology Partners Leawood /ID# 255838, Leawood, Kansas
  - Equity Medical, LLC /ID# 271140, Bowling Green, Kentucky
  - Massachusetts General Hospital /ID# 261093, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 253811, Boston, Massachusetts
  - Beacon Clinical Research, LLC /ID# 254419, Quincy, Massachusetts
  - UMass Memorial Medical Center /ID# 258839, Worcester, Massachusetts
  - The Derm Institute Of West Michigan /ID# 275948, Caledonia, Michigan
  - Hamzavi Dermatology - Canton /ID# 275856, Canton, Michigan
  - Michigan Center for Medical Research /ID# 275860, Clarkston, Michigan
  - Michigan Dermatology Institute /ID# 254468, Waterford, Michigan
  - Cleaver Dermatology /ID# 254391, Kirksville, Missouri
  - Dermatology and Skin Center of Lees Summit /ID# 257546, Lee's Summit, Missouri
  - MediSearch Clinical Trials /ID# 254392, Saint Joseph, Missouri
  - SSM Health Saint Louis University Hospital /ID# 256437, St Louis, Missouri
  - Washington University School of Medicine - St. Louis /ID# 254506, St Louis, Missouri
  - Vivida Dermatology- Flamingo /ID# 254227, Las Vegas, Nevada
  - Las Vegas Dermatology /ID# 272421, Las Vegas, Nevada
  - Skin Cancer and Dermatology Institute - Reno /ID# 254410, Reno, Nevada
  - Empire Dermatology /ID# 276241, East Syracuse, New York
  - NorthWell Health - Dermatology /ID# 254704, New Hyde Park, New York
  - Schweiger Dermatology, P.C. /ID# 254232, New York, New York
  - Private Practice - Dr. Bobby Buka /ID# 276371, New York, New York
  - Onsite Clinical Solutions /ID# 254854, Charlotte, North Carolina
  - Duke University Medical Center /ID# 256898, Durham, North Carolina
  - Apex Clinical Research Center, LLC /ID# 275956, Canton, Ohio
  - ClinOhio Research Services /ID# 254851, Columbus, Ohio
  - Dermatologists of Southwest Ohio, Inc /ID# 254297, Mason, Ohio
  - Dermatology Partners - Medina /ID# 275939, Medina, Ohio
  - Lynn Institute of Oklahoma City /ID# 253791, Oklahoma City, Oklahoma
  - Oregon Health and Science University /ID# 254929, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center /ID# 254925, Hershey, Pennsylvania
  - Paddington Testing Co., Inc. /ID# 254394, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia, LLC /ID# 255308, Philadelphia, Pennsylvania
  - Medical University of South Carolina /ID# 272569, Charleston, South Carolina
  - Dermatology Associates of Knoxville /ID# 261082, Knoxville, Tennessee
  - Arlington Research Center, Inc /ID# 253805, Arlington, Texas
  - Bellaire Dermatology Associates /ID# 253797, Bellaire, Texas
  - Dermatology Treatment and Research Center /ID# 253795, Dallas, Texas
  - Modern Research Associates, PLLC /ID# 253810, Dallas, Texas
  - HRMD Research Dallas /ID# 255256, Dallas, Texas
  - Dallas Fort Worth Clinical Research Associates (DFWCRA) /ID# 256438, Grapevine, Texas
  - Suzanne Bruce and Associates-Houston /ID# 254228, Houston, Texas
  - Texas Dermatology Research Center, LLC /ID# 254928, Plano, Texas
  - Center for Clinical Studies Webster TX /ID# 254242, Webster, Texas
  - Cope Family Medicine - Ogden Clinic /ID# 276227, Bountiful, Utah
  - University of Utah /ID# 254452, Murray, Utah
  - Springville Dermatology - Springville /ID# 276225, Springville, Utah
  - University of Virginia - Dermatology /ID# 254535, Charlottesville, Virginia
  - The Education & Research Foundation, Inc. /ID# 254852, Lynchburg, Virginia
  - Virginia Clinical Research /ID# 254538, Norfolk, Virginia
  - North Sound Dermatology /ID# 254554, Mill Creek, Washington
  - Premier Clinical Research /ID# 254847, Spokane, Washington
- Argentina (7):
  - Hospital Universitario Austral /ID# 254904, Pilar, Buenos Aires
  - Buenos Aires Skin /ID# 255299, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto de Neumonologia y Dermatologia /ID# 254903, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Psoriahue Med Interdisciplinar /ID# 257202, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Consultorios Reumatologicos Pampa /ID# 255555, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Centro de Investigacion y Prevencion Cardiovascular (CIPREC) /ID# 255474, Buenos Aires
  - Hospital Italiano /ID# 254905, CABA
- Australia (5):
  - Paratus Clinical Research Woden /ID# 254670, Phillip, Australian Capital Territory
  - Momentum Clinical Research /ID# 254411, Darlinghurst, New South Wales
  - Skin Health Institute Inc /ID# 254416, Carlton, Victoria
  - Sinclair Dermatology - Melbourne /ID# 254412, East Melbourne, Victoria
  - The Alfred Hospital /ID# 254414, Melbourne, Victoria
- Austria (3):
  - Medizinische Universitaet Graz /ID# 253448, Graz, Styria
  - Duplicate_Ordensklinikum Linz GmbH Elisabethinen /ID# 253458, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 254096, Vienna, Vienna
- Belgium (7):
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 254082, Anderlecht, Brussels Capital
  - Cliniques Universitaires UCL Saint-Luc /ID# 254087, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel /ID# 254223, Jette, Brussels Capital
  - Grand Hôpital de Charleroi - Les Viviers /ID# 254091, Charleroi, Hainaut
  - UZ Gent /ID# 254090, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 254089, Leuven, Vlaams-Brabant
  - CHU de Liege /ID# 254085, Liège
- Brazil (7):
  - Instituto de Pesquisa e Ensino CLIGEDIMUNO - IPEC /ID# 254369, Macaé, Rio de Janeiro
  - Hospital Moinhos de Vento /ID# 254366, Porto Alegre, Rio Grande do Sul
  - Hospital e Maternidade Celso Pierro - PUC-Campinas /ID# 275811, Campinas, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto /ID# 254367, Ribeirão Preto, São Paulo
  - Centro de Desenvolvimento em Estudos Clinicos Brasil - CDEC /ID# 254368, São Paulo, São Paulo
  - Instituto Brasil de Pesquisa Clinica S.A - IBPClin /ID# 275810, Rio de Janeiro
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 254370, São Paulo
- Bulgaria (4):
  - Ambulatory for Specialized Medical Care-IPSMC-skin and venereal diseases /ID# 253329, Sofiya, Sofia
  - Diagnostic Consultative Centre (Dcc) - Foкus 5 /ID# 253327, Sofiya, Sofia
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 253331, Sofia
  - UMHAT Professor Stoyan Kirkovich /ID# 253328, Stara Zagora
- Canada (20):
  - Dermatology Research Institute - Blackfoot Trail /ID# 261413, Calgary, Alberta
  - Beacon Dermatology Inc /ID# 254564, Calgary, Alberta
  - Rejuvenation Dermatology - Edmonton Downtown /ID# 254715, Edmonton, Alberta
  - Alberta Dermasurgery Centre /ID# 275945, Edmonton, Alberta
  - Care Clinic - Red Deer - Taylor Drive /ID# 276063, Red Deer, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 254378, Surrey, British Columbia
  - Enverus Medical Research /ID# 254380, Surrey, British Columbia
  - Wiseman Dermatology Research /ID# 254117, Winnipeg, Manitoba
  - Karma Clinical Trials /ID# 254120, St. John's, Newfoundland and Labrador
  - LEADER Research /ID# 254379, Hamilton, Ontario
  - DermEffects /ID# 254116, London, Ontario
  - Lynderm Research Inc /ID# 254713, Markham, Ontario
  - Derm Care Clinic /ID# 276065, Mississauga, Ontario
  - Ryan Clinical Research Inc /ID# 254714, Newmarket, Ontario
  - York Dermatology Clinic & Research Centre /ID# 254115, Richmond Hill, Ontario
  - Research Toronto /ID# 255273, Toronto, Ontario
  - CHU Sainte-Justine /ID# 254118, Montreal, Quebec
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 255632, Saint-Jérôme, Quebec
  - SkinSense Dermatology /ID# 254119, Saskatoon, Saskatchewan
  - Diex Recherche Quebec Inc. /ID# 254381, Québec
- Chile (4):
  - Centro Medico Skin Med SPA /ID# 254560, Las Condes, Region Metropolitana Santiago
  - Centro Internacional de Estudios Clinicos - CIEC /ID# 254559, Santiago, Region Metropolitana Santiago
  - Clinica Dermacross /ID# 254558, Vitacura, Region Metropolitana Santiago
  - Fundacion Innovacion Cardiovascular /ID# 254561, Independencia, Santiago Metropolitan
- Colombia (4):
  - IPS Suramericana SAS - IPS Sura San Diego /ID# 255064, Medellín, Antioquia
  - Centro de Inmunología y Genética CIGE SAS /ID# 254797, Medellín, Antioquia
  - Centro Integral de Reumatología del Caribe SAS - Circaribe SAS /ID# 255278, Barranquilla, Atlántico
  - Centro de Investigacion en Reumatologia y especialidades Medicas S.A.S- CIREEM /ID# 254796, Bogotá, Cundinamarca
- Croatia (7):
  - DermaPlus - Poliklinika za dermatologiju i venerologiju /ID# 253587, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 253786, Zagreb, City of Zagreb
  - Klinika za dječje bolesti Zagreb /ID# 253588, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 254732, Zagreb, City of Zagreb
  - Specialty Hospital Medico /ID# 254731, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 253789, Split, Split-Dalmatia County
  - Naftalan - Specijalna bolnica za medicinsku rehabilitaciju /ID# 253586, Ivanić-Grad, Zagreb County
- Czechia (3):
  - Karlovarska Krajska Nemocnice - Karlovy Vary /ID# 253456, Karlovy Vary
  - Fakultni nemocnice Kralovske Vinohrady /ID# 253454, Prague
  - Duplicate_Fakultni Nemocnice v Motole /ID# 253455, Prague
- Finland (2):
  - Oulun yliopistollinen sairaala /ID# 253969, Oulu, North Ostrobothnia
  - Terveystalo Tampere /ID# 253968, Tampere, Pirkanmaa
- France (6):
  - Chu de Nice-Hopital Larchet Ii /Id# 253504, Nice, Alpes-Maritimes
  - Centre Hospitalier Universitaire de Bordeaux - Groupe Hospitalier Saint-Andre /ID# 254139, Bordeaux, Gironde
  - Polyclinique Courlancy /ID# 254680, Reims, Marne
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 254114, Nantes, Pays de la Loire Region
  - HCL - Hopital Edouard Herriot /ID# 253500, Lyon, Rhone
  - Hopital Prive d'Antony /ID# 253501, Antony, Île-de-France Region
- Germany (15):
  - Universitaetsklinikum Freiburg /ID# 275746, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 254804, Erlangen, Bavaria
  - Universitaetsklinikum Wuerzburg /ID# 275599, Würzburg, Bavaria
  - Universitaetsklinikum Frankfurt /ID# 253683, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim /ID# 275537, Bad Bentheim, Lower Saxony
  - Studienzentrum an der Hase GbR Dr. Weyergraf/Dr. Frick/Thomas Heiber /ID# 254510, Bramsche, Lower Saxony
  - Universitaetsklinikum Duesseldorf /ID# 253711, Düsseldorf, North Rhine-Westphalia
  - Universitaetsmedizin Mainz /ID# 272596, Mainz, Rhineland-Palatinate
  - HMS GmbH Zimmer /ID# 272614, Merzig, Saarland
  - Havelklinik /ID# 254194, Berlin
  - Klinikum Ruhr Univ Bochum /ID# 253690, Bochum
  - Magdeburger Company for Medical Studies & Services GmbH /ID# 255151, Magdeburg
  - Dermatologie Quist-BAG Dres. med. Quist PartG /ID# 253691, Mainz
  - Klinik am Biederstein /ID# 254195, Munich
  - Universitaetsklinikum Regensburg /ID# 253692, Regensburg
- Greece (5):
  - 401 GSNA - 401 Army General Hospital /ID# 253499, Athens, Attica
  - University General Hospital Attikon /ID# 253495, Athens, Attica
  - General Hospital Andreas Syggros /ID# 253498, Athens, Attica
  - Hospital of Skin and Venereal Diseases- Thessaloniki /ID# 253497, Thessaloniki
  - Papageorgiou General Hospital /ID# 253496, Thessaloniki
- Hungary (9):
  - Pecsi Tudomanyegyetem Klinikai Kozpont /ID# 253753, Pécs, Baranya
  - Debreceni Egyetem-Klinikai Kozpont /ID# 253637, Debrecen, Hajdú-Bihar
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 253913, Kaposvár, Somogy County
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 254377, Szombathely, Vas County
  - Csalogany Orvosi Kozpont /ID# 255063, Budapest
  - Duplicate_Obudai Egeszsegugyi Centrum Kft. /ID# 256366, Budapest
  - Semmelweis Egyetem /ID# 276162, Budapest
  - DERMA-B Egeszsegugyi es Szolgaltato - Debrecen - Gyepusor Utca /ID# 253638, Debrecen
  - Szegedi Tudomanyegyetem /ID# 255142, Szeged
- Ireland (5):
  - St James Hospital /ID# 253973, Dublin, Dublin
  - South Infirmary Victoria University Hospital /ID# 253975, Cork
  - University College Dublin /ID# 253971, Dublin
  - University Hospital Galway /ID# 253976, Galway
  - Waterford Regional Hospital /ID# 254038, Waterford
- Israel (5):
  - ZIV Medical Center /ID# 254403, Safed, Northern District
  - Sheba Medical Center /ID# 254545, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 254404, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 254406, Haifa
  - Rabin Medical Center /ID# 254405, Petah Tikva
- Italy (9):
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale S.Anna /ID# 254496, Cona, Ferrara
  - AZIENDA USL TOSCANA CENTRO - Ospedale Piero Palagi /ID# 254495, Florence, Firenze
  - ASL 1 Abruzzo - Ospedale regionale San Salvatore /ID# 276045, L’Aquila, L Aquila
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 254498, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 254500, Rome, Roma
  - ASST degli Spedali Civili di Brescia /ID# 254875, Brescia
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 254502, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 254874, Modena
  - Azienda Ospedaliero Universitaria Pisana /ID# 254501, Pisa
- Japan (10):
  - Fukuoka University Hospital /ID# 254729, Fukuoka, Fukuoka
  - Meiwa Hospital /ID# 254728, Nishinomiya-shi, Hyōgo
  - University of Tsukuba Hospital /ID# 254638, Tsukuba, Ibaraki
  - University Hospital Kyoto Prefectural University of Medicine /ID# 254481, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 254598, Sendai, Miyagi
  - University of the Ryukyus Hospital /ID# 254517, Ginowan-shi, Okinawa
  - Kindai University Hospital /ID# 254574, Sakai, Osaka
  - Shiga University of Medical Science Hospital /ID# 254215, Ōtsu, Shiga
  - Nihon University Itabashi Hospital /ID# 254637, Itabashi-ku, Tokyo
  - Toranomon Hospital /ID# 253819, Minato-ku, Tokyo
- Lithuania (2):
  - Inlita - Santara KTC /ID# 253917, Vilnius
  - Vilnius University Hospital Santaros Klinikos /ID# 253916, Vilnius
- Mexico (3):
  - Grupo Clinico Catei Sociedad Civil /Id# 254657, Guadalajara, Jalisco
  - Eukarya PharmaSite, SC /ID# 254658, Monterrey, Nuevo León
  - Cryptex Investigacion Clinica S.A de C.V /ID# 256066, Mexico City
- Netherlands (2):
  - Amphia Ziekenhuis /ID# 253567, Breda, North Brabant
  - Universitair Medisch Centrum Groningen /ID# 253571, Groningen
- New Zealand (2):
  - Greenlane Clinical Centre /ID# 254351, Epsom, Auckland
  - Clinical Trials New Zealand /ID# 254352, Hamilton, Waikato Region
- Portugal (4):
  - Centro Hospitalar de Lisboa Central /ID# 254325, Lisbon
  - Hospital CUF Descobertas /ID# 254323, Lisbon
  - Centro Hospitalar Universitario do Porto, EPE - Hospital Santo Antonio /ID# 254322, Porto
  - Unidade Local de Saude Sao Joao, EPE /ID# 254324, Porto
- Puerto Rico (2):
  - Dr. Samuel Sanchez PSC /ID# 253948, Caguas
  - Alma M. Cruz Santana, MD-Private practice /ID# 253951, Carolina
- Saudi Arabia (4):
  - King Faisal Specialist Hospital /ID# 255539, Jeddah, Mecca Region
  - King Faisal Specialist Hospital and Research Centre /ID# 255279, Riyadh, Riyadh Region
  - King Abdulaziz Medical City- National Guard Hospital /ID# 255280, Riyadh, Riyadh Region
  - King Saud University Med City /ID# 255282, Riyadh
- Singapore (2):
  - National Skin Centre /ID# 255242, Singapore, Central Singapore
  - National University Hospital /ID# 254943, Singapore
- Slovakia (5):
  - Univerzitná nemocnica Bratislava - Nemocnica Ružinov /ID# 254157, Bratislava, Bratislava Region
  - Univerzitna nemocnica L. Pasteura Kosice /ID# 254136, Košice, Košice Region
  - Fakultna nemocnica s poliklinikou Nove Zamky /ID# 254155, Nové Zámky, Nitra Region
  - Fakultna nemocnica Trnava /ID# 254137, Trnava
  - Univerzitna nemocnica Martin /ID# 254153, Martin, Žilina Region
- South Korea (5):
  - Korea University Ansan Hospital /ID# 254128, Ansan-si, Gyeonggido
  - CHA Bundang Medical Center /ID# 254026, Seongnam, Gyeonggido
  - Seoul National University Hospital /ID# 254027, Seoul, Seoul Teugbyeolsi
  - SoonChunHyang University Seoul Hospital /ID# 254025, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital /ID# 254127, Seoul, Seoul Teugbyeolsi
- Spain (8):
  - Hospital Universitari de Bellvitge /ID# 254982, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 253924, Majadahonda, Madrid
  - Hospital de Manises /ID# 253867, Manises, Valencia
  - Hospital Santa Creu i Sant Pau /ID# 253869, Barcelona
  - Hospital General de Granollers /ID# 253873, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 253870, Granada
  - Hospital Universitario Ramon y Cajal /ID# 253871, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 253868, Valencia
- Sweden (2):
  - Karolinska University Hospital Solna /ID# 254808, Solna, Stockholm County
  - Sahlgrenska Universitetssjukhuset /ID# 254807, Gothenburg, Västra Götaland County
- Switzerland (3):
  - Kantonsspital St. Gallen /ID# 255243, Sankt Gallen, Canton of St. Gallen
  - University Hospital Zurich /ID# 254642, Zurich, Canton of Zurich
  - Inselspital, Universitaetsspital Bern /ID# 254736, Bern
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 254031, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 254030, Taipei City, Taipei
  - Changhua Christian Hospital /ID# 254032, Changhua City, Changhua County
  - Linkou Chang Gung Memorial Hospital /ID# 254033, Taoyuan
- Turkey (Türkiye) (6):
  - Gulhane Egitim ve Arastirma Hastanesi /ID# 253919, Ankara, Antalya
  - Izmir Sehir Hastanesi /ID# 265465, Bayraklı
  - Uludag University Medical Faculty /ID# 253806, Bursa
  - Istanbul Universitesi-Cerrahpasa Cerrahpasa Tip Fakultesi /ID# 253824, Istanbul
  - Erciyes University Medical Faculty /ID# 253804, Kayseri
  - Ondokuz Mayis Universitesi /ID# 254034, Samsun
- United Kingdom (7):
  - Chelsea and Westminster Hospital /ID# 254190, London, Greater London
  - St George University Hospitals NHS Foundation Trust /ID# 256803, London, Greater London
  - University Hospital Southampton NHS Foundation Trust /ID# 254531, Southampton, Hampshire
  - UH Coventry & Warwickshire /ID# 256909, Coventry, Warwickshire
  - Leeds Teaching Hospitals NHS Trust /ID# 254616, Leeds, West Yorkshire
  - University Hospitals Bristol /ID# 261505, Bristol
  - Northern Care Alliance NHS Group /ID# 256910, Salford

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-698